CLINICAL TRIAL: NCT02326649
Title: Noninvasive Measurement of Cardiac Output Using Impedance Cardiography in Patients With Congenital Heart Disease
Brief Title: Noninvasive Measurement of CO Using Impedance Cardiography in Patients With CHD
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dr. Christopher Davis, PI, University of California, San Diego
Other Study IDs: 140550
Record Dates: First submitted 2014-12-15; First posted 2014-12-29 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-02

CONDITIONS: Congenital Heart Disease
Keywords: cardiac output
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHD patients undergoing cardiac MRI without sedation
  Interventions: Device: Physioflow

INTERVENTIONS:
Device: Physioflow — impedance cardiography instrument that measures cardiac output non-invasively

SUMMARY:
This study will test the capability of a non-invasive instrument (the PhysioFlow impedance cardiography instrument) to measure cardiac output in patients with congenital heart disease (CHD). This instrument works by placing electrodes on the skin of a patient and measuring electrical impedance through the chest, which is proportional to blood volume and blood flow at any given time. The instrument has been validated in patients with structurally normal hearts, but in the only two studies using it for patients with CHD, it was deemed too inaccurate for clinical use. The manufacturer of the device would require access to data on the patients in order to improve its accuracy, and that has not been feasible thus far. This study would begin by comparing cardiac output based on the PhysioFlow monitor to standard techniques, then after possible changes to the instrument to enhance accuracy, would test the instrument again in the same way.

DETAILED DESCRIPTION:
The measurement of cardiac output (CO) is important for a wide variety of patients under multiple conditions. At present, gold standard techniques for measurement of CO include velocity encoded phase contrast MRI. Both of these techniques are valid in patients with structural CHD. Disadvantages of these techniques include the requirement of significant time and expertise, and the high cost and anesthesia requirement. Accurate, non-invasive tools to measure CO could be extremely valuable for patients with CHD that require one-time of continuous monitoring of CO, such as during surgery, in intensive care settings, during other diagnostic testing, and during different physiologic states such as sleep and exercise. This study would begin by comparing cardiac output based on the PhysioFlow monitor to cardiac outout by MRI.

Impedance cardiography is performed by placing electrodes on the thorax and neck to measure electrical impedance over time. Cardiac output is derived from these measurements. The technique has been studied, validated, and used extensively in adults and has also been shown to be valid in children with structurally normal hearts. In contrast, recent studies of children with CHD have shown a relatively poor agreement between impedance cardiography and both thermodilution technique and velocity encoded phase contrast MRI. The reasons for the poor agreement in CHD patients is not yet understood. There are proprietary algorithms in each impedance device that use the raw data to calculate and report cardiac output. If the physiologic and/or anatomic differences of patients with CHD require changing the algorithm within each system to account for such differences, that needs to be done to each system. In order to do this, owners of any given device (PhysioFlow, NeuMeDx Inc. in this case) need access to the raw data in order to alter the algorithm. This study will involve a concerted effort between investigators at RCHSD, UCSD, and NeuMeDx

ELIGIBILITY:
Inclusion Criteria:

* Any form of congenital heart disease
* Any age

Exclusion Criteria:

* Subjects with significant clinical skin reactions to electrodes such as excessive pain and/or skin inflammation, or significant previous skin reaction
* Subjects who are not able to provide consent
* Subjects with pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with congenital heart disease that is undergoing cardiac MRI without anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SMIC and CMR: Participants with various congenital heart disease diagnoses with both signal-morphology IC (SMIC) measurements and cardiac magnetic resonance (CMR) imaging
Period: Overall Study
Arm/Group | SMIC and CMR
Started | 33
Completed | 21
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Diagnosis, Age, and Body Size of Subjects: Overall
Arm/Group | Diagnosis, Age, and Body Size of Subjects
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 18 [7 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Surface Area [Mean (Full Range); unit: meters squared] | 1.67 [0.8 to 2.2]

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Stroke Volume Between CMR and SMIC
Description: Mean difference in stroke volume (SV) between CMR and SMIC measurements in ml
Time Frame: 2 hours
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | SMIC and CMR
Number analyzed (Participants) | 21
ml | 1.7 [-3.1 to 6.6]
Statistical Analysis 1: Comparison: SMIC and CMR; Test type: Other; p = 0.47, paired t-test
Statistical Analysis 2: Comparison: SMIC and CMR; Intercept for multilinear regression for difference in stroke volume controlling for difference in heart rate and blood pressure; Test type: Other; p = 0.255, Regression, Linear; Mean Difference (Final Values) = 6.561, 95% CI 2-sided [-5.295 to 18.417], Standard Error of Mean 5.528
Statistical Analysis 3: Comparison: SMIC and CMR; Heart rate delta for multilinear regression for difference in stroke volume controlling for difference in heart rate and blood pressure; Test type: Other; p = 0.250, Regression, Linear; Mean Difference (Final Values) = 0.500, 95% CI 2-sided [-0.395 to 1.395], Standard Error of Mean 0.417
Statistical Analysis 4: Comparison: SMIC and CMR; Diastolic BP delta for multilinear regression for difference in stroke volume controlling for difference in heart rate and blood pressure; Test type: Other; p = 0.183, Regression, Linear; Mean Difference (Final Values) = -0.427, 95% CI 2-sided [-1.081 to 0.227], Standard Error of Mean 0.305
Statistical Analysis 5: Comparison: SMIC and CMR; Systolic BP delta for multilinear regression for difference in stroke volume controlling for difference in heart rate and blood pressure; Test type: Other; p = 0.238, Regression, Linear; Mean Difference (Final Values) = 0.557, 95% CI 2-sided [-0.411 to 1.526], Standard Error of Mean 0.452

ADVERSE EVENTS:
Arm/Group | CHD Patients Undergoing Cardiac MRI Without Sedation
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No